CLINICAL TRIAL: NCT00860171
Title: A Study Evaluating Escalating Doses of 131I-BC8 (Anti-CD45) Antibody Followed by Autologous Stem Cell Transplantation for Relapsed or Refractory Lymphoid Malignancies
Brief Title: Iodine I 131 Monoclonal Antibody BC8 Before Autologous Stem Cell Transplant in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma or Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to lack of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2238.00; NCI-2010-00128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2238.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2019-08

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Hodgkin Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Hodgkin Disease; Lymphoma, T-Cell | interventions — Iodine-131

STUDY DESIGN:
Intervention Model Description: A single site, open label clinical trial.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (iodine I 131 monoclonal antibody B, autologous HCT) (Experimental): Patients receive a dosimetric dose of iodine I 131 monoclonal antibody BC8 IV on day -20 and a therapeutic dose on day -11. Before day -20, patients may also receive up to 2 additional dosimetric doses of iodine I 131 monoclonal antibody BC8 IV approximately 1-2 weeks apart. Patients then undergo autologous stem cell transplantation on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Radiation: Iodine I 131 Monoclonal Antibody BC8; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Autologous stem cells given via central catheter
  Other Names: Autologous Stem Cell Transplantation
Radiation: Iodine I 131 Monoclonal Antibody BC8 — Given IV
  Other Names: I 131 MOAB BC8; I 131 Monoclonal Antibody BC8; iodine I 131 MOAB BC8; MOAB BC8, iodine I 131; monoclonal antibody BC8, iodine I 131
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of iodine I 131 monoclonal antibody BC8 when given before autologous stem cell transplant in treating patients with Hodgkin lymphoma or non-Hodgkin lymphoma that has returned after a period of improvement or does not respond to treatment. Radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving iodine I 131 monoclonal antibody BC8 before an autologous stem cell transplant may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximally tolerated dose of 131I-BC8 (anti-cluster of differentiation [CD]45) (iodine I 131 monoclonal antibody BC8) that can be delivered prior to autologous stem cell transplantation for patients with relapsed/refractory B-non-Hodgkin lymphoma (NHL), T-NHL, or Hodgkin lymphoma (HL).

SECONDARY OBJECTIVES:

I. To optimize the protein dose (antibody [Ab]) to deliver a favorable biodistribution in the majority of patients.

II. To assess the radiation dose delivered to tumor sites and normal organs by the above therapy.

III. To evaluate the dose-response relationship of radiation-dose to tumor and clinical response.

IV. To estimate the overall and progression-free survival of the above regimen in such patients.

V. To evaluate the toxicity and tolerability of the above therapy.

VI. To evaluate the feasibility of delivering high-dose 131I-BC8 and autologous stem cell transplantation (ASCT) to B-Cell NHL, T-NHL, and HL patients.

VII. To evaluate the ability to reduce infusion reactions via unlabeled BC8 preinfusion.

OUTLINE: This is a dose-escalation study.

Patients receive a dosimetric dose of iodine I 131 monoclonal antibody BC8 intravenously (IV) on day -20 and a therapeutic dose on day -11. Before day -20, patients may also receive up to 2 additional dosimetric doses of iodine I 131 monoclonal antibody BC8 IV approximately 1-2 weeks apart. Patients then undergo autologous stem cell transplantation on day 0.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of B-NHL, T-NHL, or HL; CD45 antigen expression must be documented on tumor specimens in all cases except HL, in whom histologic demonstration of CD45+ cells adjacent to the Reed Sternberg cells is required
* Patients must have received at least one prior standard systemic therapy with documented recurrent or refractory disease
* Mantle cell lymphoma (MCL), T-NHL, or other high-risk malignancies may be enrolled/transplanted in complete remission (CR)/first partial remission (PR1)
* Patients are preferred to have either a tumor mass amenable to core needle biopsy during the dosimetry phase, or a measurable tumor mass with at least one site of involvement measuring 2.0 cm in largest dimension on computed tomography (CT) imaging for purposes of planar and/or single-photon emission CT (SPECT)/CT tumor dosimetry (patients with disease that does not allow tumor dosimetry will be allowed on study since they still can contribute toward achieving the primary endpoint, but these patients will be given a lower priority over those with evaluable disease)
* Creatinine [Cr] < 2.0
* Bilirubin < 1.5 mg/dL, with the exception of patients thought to have Gilbert's syndrome, who may have a total bilirubin above 1.5 mg/dL
* All patients eligible for therapeutic study must have a minimum of >= 4 x10^6 CD34/kg autologous hematopoietic stem cells harvested and cryopreserved and divided into 2 aliquots of at least >= 2 x10^6 CD34/kg each; patients with a history of prior autologous hematopoietic cell transplant (HCT) are only required to have >= 2x10^6 CD34/kg stored
* Patients must have an expected survival of > 60 days and must be free of major infection

Exclusion Criteria:

* Circulating human anti-mouse antibody (HAMA), to be determined before each infusion
* Systemic anti-lymphoma therapy given in the previous 30 days before the scheduled therapy dose with the exception of rituximab
* Inability to understand or give an informed consent
* Lymphoma involving the central nervous system
* Other serious medical conditions considered to represent contraindications to bone marrow transplant (BMT) (e.g. abnormally decreased cardiac ejection fraction, diffusion capacity of the lung for carbon monoxide (DLCO) < 50% predicted, forced expiratory volume in one second (FEV1) < 70% predicted, acquired immune deficiency syndrome [AIDS], etc.)
* Known human immunodeficiency virus (HIV) seropositivity
* Pregnancy or breast feeding
* Prior allogeneic bone marrow or stem cell transplant
* Prior autologous bone marrow or stem cell transplant or prior radiation therapy (RT) > 20 Gy to a critical organ within 1 year of enrollment
* Presence of circulating lymphoma cells by morphology or flow cytometry (> 0.1%) at or near the time of peripheral blood stem cell (PBSC) collection if unpurged/unselected PBSC are to be used (patients with cryopreserved stem cells which are negative [=< 0.1% involved] by flow cytometry will also be considered eligible)
* Southwest Oncology Group (SWOG) performance status >= 2.0
* Unable to perform self-care during radiation isolation
* Expected survival if untreated less than 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2015-03 (Actual); Study Completion 2020-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.81 (15.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of I-131-BC8 That Can be Delivered Prior to Transplant
Description: Dose escalation/de-escalation will be conducted by the "two-stage" approach introduced by Storer. Escalation will continue until a dose-limiting toxicity (DLT) occurs. A DLT will be defined as a therapy-related grade III or IV Bearman (transplant) toxicity. The MTD is estimated to be the dose that is associated with a toxicity rate of 25% (Bearman grade 3-4).
Time Frame: Within 30 days post-transplant
Measure: Number; unit: Gray of I-131 (absorbed dose that the I
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
Gray of I-131 (absorbed dose that the I | NA — No dose-limiting toxicities observed. Funding ran out, and no MTD identified by the time last patient treated.

2. Primary Outcome: I-131 Activity Administered
Time Frame: At time of I-131 therapy
Measure: Mean (Full Range); unit: mCi I-131
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
mCi I-131 | 668.15 [344 to 1064]

3. Secondary Outcome: Adverse Events
Description: Descriptive statistics will be calculated. DLT will be defined by the Bearman Scale that is designed to address the specific toxicities associated with transplantation.
Time Frame: Up to 6 years
Measure: Number; unit: number of adverse events
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
number of adverse events | 0

4. Secondary Outcome: Overall Survival
Time Frame: Up to 6 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
days | 1057 (633.59)

5. Secondary Outcome: Progression-free Survival
Description: number of people with progression free survival
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
Participants | 5

6. Secondary Outcome: Relapse Rate
Description: Number of relapse
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Number analyzed (Participants) | 16
Participants | 5

ADVERSE EVENTS:
Arm/Group | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT)
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Iodine I 131 Monoclonal Antibody B, Autologous HCT) (N=16)
Fever (General disorders) | 1 (1) — non-neutropenic fever
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This protocol was closed to enrollment when replaced by a newer approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes